CLINICAL TRIAL: NCT01906476
Title: Stepped Telemental Health Care Intervention for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Mohr, Director, Center for Behavioral Intervention Technologies; Professor, Department of Preventive Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH095753-01A1-RCTTH; R01MH095753-01A1 (NIH)
Record Dates: First submitted 2013-07-17; First posted 2013-07-24 (Estimated); Results first posted 2020-04-02 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Depression
Keywords: Depression; Telephone Cognitive Behavior Therapy; Internet Cognitive Behavioral Therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stepped Care (Experimental): Participants will receive an Internet guided cognitive behavioral treatment (iCBT) with support from a telephone coach with the possibility of being stepped up to receiving telephone cognitive behavior therapy (T-CBT) with a therapist
  Interventions: Behavioral: Stepped Care
- Telephone Cognitive Behavior Therapy (Active Comparator): Participants will receive telephone-administered cognitive behavioral therapy (T-CBT).
  Interventions: Behavioral: Telephone Cognitive Behavior Therapy

INTERVENTIONS:
Behavioral: Stepped Care — Participants will receive an Internet guided cognitive behavioral treatment (iCBT) with support from a telephone coach with the possibility of being stepped up to receiving telephone cognitive behavior therapy (T-CBT) with a therapist
  Arms: Stepped Care
Behavioral: Telephone Cognitive Behavior Therapy — Participants will receive telephone-administered cognitive behavioral therapy (T-CBT).
  Arms: Telephone Cognitive Behavior Therapy

SUMMARY:
This is a randomized, controlled trial comparing telephone-cognitive behavior therapy (T-CBT) with a therapist to a "Stepped Care" intervention for depression treatment (iCBT with support from a telephone coach with the possibility of being stepped up to receiving T-CBT with a therapist).

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is common, with 12-month prevalence rates estimated to be between 6.6-10.3%. While many depressed patients state they would prefer psychological treatment to pharmacotherapy, substantial barriers to care exist, including cost, practical barriers such as time constraints and transportation, emotional barriers such as stigma, decreased motivation associated with depression itself, physical disability, and lack of availability of services. Telemental health has been proposed as a method of overcoming barriers to treatment. Research has focused primarily on two formats: the telephone and the Internet. Use of the telephone as a delivery medium produces reductions in depression equivalent to face-to-face psychological treatments, while also significantly reducing attrition. However, its success in outreach can also significantly increase costs for healthcare providing organizations. Internet interventions have the potential to produce moderate gains when supported by therapist or coach via brief telephone calls or e-mail but are also less expensive than standard therapy. Developing healthcare models that integrate treatment delivery media holds the promise of harnessing the advantages of each media, while minimizing the disadvantages. Stepped care models are a potentially useful framework for achieving such an integration. The stepped care model we will test initiates treatment with a validated, guided Internet cognitive behavioral therapy program. If patients fail to respond, they will be stepped up to a validated telephone-cognitive behavior therapy (T-CBT). The stepped care model will be compared to T-CBT in a randomized trial. Patients will be recruited from primary care and treated for up to 20 weeks, or until sustained remission is achieved.

ELIGIBILITY:
Inclusion Criteria:

* Has a DSM-IV diagnosis of non-psychotic major depressive disorder (MDD) as assessed using the Mini International Neuropsychiatric Interview (MINI), plus a score of 12 or greater on the Quick Inventory of Depressive Symptomatology - Clinician Rated (QIDS-C)
* Has a phone, access to the Internet, and basic internet skills
* Is at least 18 years of age
* Is able to speak and read English
* If currently taking an antidepressant medication, participant must have been on a stable dose for at least two weeks, and have no plans to change the dose

Exclusion Criteria:

* Has visual, hearing, voice, or motor impairment that would prevent completion of study procedures
* Is diagnosed with a psychotic disorder, bipolar disorder, dissociative disorder, substance use or other diagnosis for which participation in this trial is either inappropriate or dangerous
* Is severely suicidal (has ideation, plan, and intent)
* Is currently receiving or planning to begin psychotherapy during the study treatment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Mohr, Ph.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohr DC, Lattie EG, Tomasino KN, Kwasny MJ, Kaiser SM, Gray EL, Alam N, Jordan N, Schueller SM. A randomized noninferiority trial evaluating remotely-delivered stepped care for depression using internet cognitive behavioral therapy (CBT) and telephone CBT. Behav Res Ther. 2019 Dec;123:103485. doi: 10.1016/j.brat.2019.103485. Epub 2019 Sep 30. PMID 31634738

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stepped Care | Telephone Cognitive Behavior Therapy
Started | 157 | 155
Completed | 140 | 139
Not Completed | 17 | 16
Not completed — Lost to Follow-up | 17 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stepped Care | Telephone Cognitive Behavior Therapy | Total
Number analyzed (Participants) | 157 | 155 | 312
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [27 to 49] | 32 [26 to 45.5] | 33 [27 to 47]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two patients did not report their gender.
  Participants
    number analyzed (Participants) | 155 | 155 | 310
    Female | 118 | 111 | 229
    Male | 37 | 44 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 20 | 32
  Not Hispanic or Latino | 141 | 134 | 275
  Unknown or Not Reported | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 5 | 6 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 9 | 14
  White | 135 | 130 | 265
  More than one race | 7 | 5 | 12
  Unknown or Not Reported | 5 | 3 | 8
Baseline QIDS (Quick Inventory of Depressive Symptomatology) [Median (Inter-Quartile Range); unit: units on a scale] — QIDS is made up of 16 items and has a possible range of scores of 0 to 27. Higher scores represent worse outcomes.
  units on a scale | 14 [13 to 16] | 14 [13 to 17] | 14 [13 to 16.25]
PHQ-9 (Patient Health Questionnaire 9) [Median (Inter-Quartile Range); unit: units on a scale] — PHQ-9 is made up of 9 items and has a possible range of scores of 0 to 27. Higher scores represent worse outcomes.
  units on a scale | 16 [14 to 19] | 17 [14 to 19] | 16 [14 to 19]

OUTCOME MEASURES:

1. Primary Outcome: Depression
Description: To measure changes in the Quick Inventory of Depressive Symptomatology (QIDS) over time. The QIDS is made up of 16 items and has a possible range of scores of 0 to 27. Higher scores represent worse outcomes.
Time Frame: Baseline, midtreatment, end of treatment, 3 month post treatment, and 6 month post-treatment follow-up
Population: Participants with at least one followup visit which recorded the QIDS post baseline
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Stepped Care | Telephone Cognitive Behavior Therapy
Number analyzed (Participants) | 134 | 136
units on a scale
  Midtreatment | 10.51 (0.40) | 11.22 (0.39)
  End of Treatment | 7.84 (0.38) | 7.71 (0.37)
  Month 3 (post treatment) | 7.78 (0.42) | 7.88 (0.40)
  Month 6 (post treatment) | 7.89 (0.44) | 8.24 (0.42)
Statistical Analysis 1: Comparison: Stepped Care vs Telephone Cognitive Behavior Therapy; Test type: Non-Inferiority — Non-inferiority trials of pharmaceuticals have used 30% to 50% of the difference between treatment and control conditions to define non-inferiority margins. (Jones, Jarvis, Lewis, & Ebbutt, 1996; Nutt et al., 2008). A meta-analysis of CBT found an overall effect size of d=0.82.(Cuijpers, Smit, Bohlmeijer, Hollon, & Andersson, 2010). Using the midpoint of 40% for the acceptable criterion, we set d=0.33 as the non-inferiority criterion; Cohen's d and upper limits of one-sided 95% Confidence intervals for each time are as follows: Mid-treatment -0.19 (95% upper limit= 0.06) End of treatment 0.03 (0.24) 3 months post treatment -0.02 (0.19) 6 months post treatment -0.07 (0.14)

2. Primary Outcome: Cost-Effectiveness
Description: Measure the ratio of the difference in costs and difference in effectiveness between the two groups, Stepped care minus Telephone Cognitive Behavior Therapy. Below are reported individual cost means and standard deviations for therapist costs during study.
Time Frame: Baseline to end of treatment
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Stepped Care | Telephone Cognitive Behavior Therapy
Number analyzed (Participants) | 157 | 155
dollars | 391.81 (229.06) | 756.14 (298.64)
Statistical Analysis 1: Comparison: Stepped Care vs Telephone Cognitive Behavior Therapy; We calculated the ICER (Incremental cost-effectiveness ratio) estimate, computed using the difference in average cost between the two arms, divided by the difference in average Depression Free Days (DFD) as defined using QIDS (Quick Inventory of Depressive Symptomatology), between the two arms, Stepped Care minus Telephone Cognitive Behavior Therapy. The confidence interval was created using bootstrapping; Test type: Superiority; ICER estimate = -152.55, 95% CI 2-sided [-1143.09 to 1094.72]

ADVERSE EVENTS:
Time Frame: Baseline through 6 month post-treatment followup
Arm/Group | Stepped Care | Telephone Cognitive Behavior Therapy
All-Cause Mortality (participants affected / at risk) | 0/157 | 0/155
Serious Adverse Events (participants affected / at risk) | 0/157 | 0/155
Other Adverse Events (participants affected / at risk) | 0/157 | 0/155

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT01906476/Prot_SAP_000.pdf